CLINICAL TRIAL: NCT02700126
Title: Impact of Genetic Polymorphism on Propofol Requirement and Recovery for Total Intravenous Anesthesia for Clipping of Unruptured Cerebral Aneurysm in Korean Population
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-1195
Record Dates: First submitted 2016-02-26; First posted 2016-03-07 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Unruptured Cerebral Aneurysm
Keywords: propofol; total intravenous anesthesia; cerebral aneurysm; single nucleotide polymorphism
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood obtained from enrolled patients before surgery
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- undergoing propofol based TIVA for clip: This study is an observational study performed in adult patients undergoing propofol based TIVA for clipping of unruptured cerebral aneurysm. We will collect data regarding recovery after stopping propofol infusion (time for eye opening and extubation), propofol requirement during anesthesia maintenance, and propofol effect site concentration to achieve bispectral index 40 during anesthesia induction, without doing any interventions. Data collection will be established with just observing and recording values displayed in screens of monitoring devices, and reviewing patient charts.

SUMMARY:
In neurosurgical anesthesia, propofol based total intravenous anesthesia (TIVA) is frequently used due to brain relaxation and less effect on electrophysiologic monitoring. Response to propofol can vary between individuals and be associated with clinical factors including age and weight, and genetic polymorphism. Because the importance of rapid recovery in neurosurgery with long operation time is emphasized recently, the choice and dose adjustment of anesthetics should be determined according to clinical and genetic factors. Recently, researches about genetic variations have been performed with single nucleotide polymorphism (SNP). The aim of this study is to determine SNPs associated with propofol recovery and response in Korean adult population undergoing propofol based TIVA for clipping of unruptured cerebral aneurysm.

ELIGIBILITY:
Inclusion Criteria:

1. Korean adult population undergoing propofol based TIVA for clipping of unruptured cerebral aneurysm

Exclusion Criteria:

1. patients not able to read, or understand the consent form
2. ethnicity, other than Korean population
3. patients refusal
4. patients not to perform total intravenous anesthesia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean adult population undergoing propofol based total intravenous anesthesia for clipping of unruptured cerebral aneurysm.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

PRIMARY OUTCOMES:
Time of eye opening after stopping propofol infusion | within about one hour from end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share data

REFERENCES:
- [Background] Iohom G, Ni Chonghaile M, O'Brien JK, Cunningham AJ, Fitzgerald DF, Shields DC. An investigation of potential genetic determinants of propofol requirements and recovery from anaesthesia. Eur J Anaesthesiol. 2007 Nov;24(11):912-9. doi: 10.1017/S0265021507000476. Epub 2007 Jun 7. PMID 17555608